CLINICAL TRIAL: NCT07231471
Title: Platelet Rich Plasma for Musculoskeletal Conditions
Acronym: PRP for MSK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Daniel Cushman, Principal Investigator, Clinical Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00191115
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis (OA); Osteoarthritis (OA) of the Knee; Osteoarthritis (OA) of the Hip; Osteoarthritis (OA) of the Shoulder; Osteoarthritis Ankle; Elbow Osteoarthritis; Epicondylitis of the Elbow; Plantar Fasciitis of Both Feet; Tendinopathy
Keywords: PRP; Platelet Rich Plasma; Osteoarthritis; Tendinopathy
MeSH Terms: conditions — Osteoarthritis; Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Platelet Rich Plasma Injection (Experimental): Participants who are eligible and provide consent to participate will undergo a Platelet-Rich Plasma (PRP) injection. Their whole blood and the produced PRP will be analyzed using a cell counter, and they will be asked to complete follow-up surveys at 2 weeks, 6 weeks, 3 months, 6 months, and 12 months..
  Interventions: Biological: Platelet Rich Plasma Injection; Device: Platelet Rich Plasma Preparation

INTERVENTIONS:
Biological: Platelet Rich Plasma Injection — Participants who are eligible and provide consent to participate will undergo a Platelet-Rich Plasma (PRP) injection. Their blood will be analyzed using a cell counter, and they will be asked to complete follow-up surveys at 2 weeks, 6 weeks, 3 months, 6 months, and 12 months.
Device: Platelet Rich Plasma Preparation — The patient's blood is collected into syringes. That blood is spun in a centrifuge at high speeds, which separates their blood into layers (red blood cells, white blood cells, and plasma). The plasma portion, which contains the platelets, is transferred to a different syringe for later injection. In some cases, the plasma is spun in the centrifuge again (a "double spin" technique) to further concentrate the platelets in the plasma. The patient's blood is not exposed to air, and it is transferred by tubing between syringes with a Luer Lock connection.

SUMMARY:
The primary purpose of this study is to follow patients with various musculoskeletal (MSK) conditions over a one-year follow-up period after receiving a platelet rich plasma (PRP) injection, assessing changes in their pain levels, functional abilities, and overall patient satisfaction.

This will develop a robust registry of patients treated with PRP for a range of MSK conditions. These conditions include, but are not limited to, osteoarthritis (OA) of the knee, hip, glenohumeral joint, elbow, ankle, and sacroiliac joint, as well as rotator cuff tendinopathy, lateral and medial epicondylitis, plantar fasciitis, patellar tendinopathy, Achilles tendinopathy, and proximal hamstring tendinopathy.

DETAILED DESCRIPTION:
Platelet-Rich Plasma (PRP) is an injectable preparation of a patient's blood that can be used for numerous conditions and has received significant attention over the past several years for its potential application for the treatment of pain and functional impairment due to osteoarthritis (OA) and other musculoskeletal conditions. Research on PRP has expanded dramatically over the last several decades, elevating its status from snake oil to a proven injection option superior to corticosteroids. It has demonstrated superior efficacy to standard-of-care corticosteroids in numerous musculoskeletal conditions. Systematic reviews of randomized-controlled trials have demonstrated equivalent-to-superior treatment outcomes associated with the use of intra-articular PRP compared to placebo, hyaluronic acid, and corticosteroid for the most commonly-studied condition, knee OA. Most importantly, just as corticosteroids have been used in numerous musculoskeletal conditions (OA, tendinopathy, bursitis, etc.), PRP has the same potential, but with vastly reduced risk; corticosteroids have many known dangers. To summarize, PRP has demonstrated level 1 evidence of superiority to corticosteroids in pain and function in numerous musculoskeletal conditions, with considerably less risk.

This study will evaluate pain, function, and overall patient satisfaction outcomes for the use of PRP for the treatment of a diverse MSK conditions, including, but not limited to, OA of the knee, hip, glenohumeral joint, elbow, ankle, and sacroiliac joint, as well as rotator cuff tendinopathy, lateral and medial epicondylitis, plantar fasciitis, patellar tendinopathy, Achilles tendinopathy, and proximal hamstring tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Musculoskeletal pathology that may benefit from a PRP injection
* Failed other conservative treatments

Exclusion Criteria:

* No active malignancy
* No active infection in the area of injection
* No platelet disorder
* No active systemic infections
* No patients currently undergoing dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog score (pain) | 6 months
  The VAS is a 0 to 10 scale, with zero being no pain and ten being the worst pain imaginable for their condition

SECONDARY OUTCOMES:
Visual Analog Score (pain) | 1, 3, and 12 months
  The VAS is a 0 to 10 scale, with zero being no pain and ten being the worst pain imaginable for their condition
Global satisfaction | 1, 3, 6, 12 months
  From a scale of 0 to 100, the subject assesses their total satisfaction with the affected body part. Zero is no satisfaction, while 100 is complete satisfaction.
Western Ontario and McMaster Universities Arthritis Index (knee) | 1, 3, 6, 12 months
  The WOMAC is a self-administered questionnaire used to evaluate pain, stiffness, and physical function in people with hip and knee osteoarthritis. Only for patients with knee OA.
  WOMAC scoring involves summing the scores from its three subscales: pain (5 items), stiffness (2 items), and physical function (17 items). Each subscale has a maximum score (Pain: 20, Stiffness: 8, Physical Function: 68), and a total WOMAC score is calculated by adding these three sub-scores together, for a possible total range of 0-96. Higher scores indicate worse symptoms and function.
Disorders of the Arm, Shoulder, and Hand (QuickDASH) | 1, 3, 6, 12 months
  The QuickDASH an 11-item patient-reported questionnaire used to measure physical function and symptoms in people with musculoskeletal disorders of the upper limb (arm, shoulder, and hand).
  To score the QuickDASH, the first sum is the scores from the 11 items, each rated on a 1-5 Likert scale.
  The sum is then used in the formula: QuickDASH Score = ([(sum of n responses)/n]-1)*25), where (n) is the number of completed items. A minimum of 10 out of 11 items must be completed to calculate a score, and the final score ranges from 0 (no disability) to 100 (most severe disability).
International Hip Outcome Tool 12 (IHOT12) | 1, 3, 6, 12 months
  This is a 12-item patient-reported outcome measure (PROM) used to assess the health-related quality of life in young, active patients with hip problems. Each question is scored from 0 (worst symptoms/function) to 100 (best symptoms/function). The scores are averaged from all questions, and the final score ranges from 0 (worst symptoms/function) to 100 (best symptoms/function).
Foot and Ankle Outcome Score (FAOS) | 1, 3, 6, 12 months
  The FAOS is a patient-reported questionnaire that measures a person's foot and ankle symptoms and functional status. It is divided into five subscales: pain, other symptoms, function in daily living, function in sports and recreation, and quality of life. Scores for each subscale range from 0 to 100, where 100 represents no symptoms and 0 indicates the worst possible symptoms.
EQ-5D | 1, 3, 6, 12 months
  The EQ-5D is a self-report questionnaire that measures health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It consists of two parts of the EURO-QOL.
  The first is an index score, calculated from a 5-digit health state code that corresponds to a person's self-reported level of problems in five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). It is calculated by applying a formula to the 5-digit descriptive system code (e.g., 11111 for no problems). This formula uses "social preference weights" for each level in each dimension. A score of 1 represents perfect health, while 0 represents death. Negative scores are possible for health states considered "worse than dead".
  The second is an EQ-VAS score, a direct self-assessment on a visual analog scale from 0 (worst imaginable health) to 100 (best imaginable health).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Orthoaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cushman DM, Johnson LA, Burnham T, Nelson R, Egbert J, Burnham R. An evaluation of a low-cost platelet-rich plasma for osteoarthritis of the knee: A pilot study. J Exp Orthop. 2025 Sep 5;12(3):e70420. doi: 10.1002/jeo2.70420. eCollection 2025 Jul. PMID 40919485
- [Background] Baria MR, Vasileff WK, Borchers J, DiBartola A, Flanigan DC, Plunkett E, Magnussen RA. Treating Knee Osteoarthritis With Platelet-Rich Plasma and Hyaluronic Acid Combination Therapy: A Systematic Review. Am J Sports Med. 2022 Jan;50(1):273-281. doi: 10.1177/0363546521998010. Epub 2021 Apr 8. PMID 33831332
- [Background] Elksnins-Finogejevs A, Vidal L, Peredistijs A. Intra-articular platelet-rich plasma vs corticosteroids in the treatment of moderate knee osteoarthritis: a single-center prospective randomized controlled study with a 1-year follow up. J Orthop Surg Res. 2020 Jul 10;15(1):257. doi: 10.1186/s13018-020-01753-z. PMID 32650801
- [Background] Forogh B, Mianehsaz E, Shoaee S, Ahadi T, Raissi GR, Sajadi S. Effect of single injection of platelet-rich plasma in comparison with corticosteroid on knee osteoarthritis: a double-blind randomized clinical trial. J Sports Med Phys Fitness. 2016 Jul-Aug;56(7-8):901-8. Epub 2015 Jul 14. PMID 26173792
- [Background] Joshi Jubert N, Rodriguez L, Reverte-Vinaixa MM, Navarro A. Platelet-Rich Plasma Injections for Advanced Knee Osteoarthritis: A Prospective, Randomized, Double-Blinded Clinical Trial. Orthop J Sports Med. 2017 Feb 13;5(2):2325967116689386. doi: 10.1177/2325967116689386. eCollection 2017 Feb. PMID 28255569
- [Background] Tan J, Chen H, Zhao L, Huang W. Platelet-Rich Plasma Versus Hyaluronic Acid in the Treatment of Knee Osteoarthritis: A Meta-analysis of 26 Randomized Controlled Trials. Arthroscopy. 2021 Jan;37(1):309-325. doi: 10.1016/j.arthro.2020.07.011. Epub 2020 Jul 15. PMID 32679294
- [Background] Habib GS. Systemic effects of intra-articular corticosteroids. Clin Rheumatol. 2009 Jul;28(7):749-56. doi: 10.1007/s10067-009-1135-x. Epub 2009 Feb 28. PMID 19252817
- [Background] Dai WL, Zhou AG, Zhang H, Zhang J. Efficacy of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Meta-analysis of Randomized Controlled Trials. Arthroscopy. 2017 Mar;33(3):659-670.e1. doi: 10.1016/j.arthro.2016.09.024. Epub 2016 Dec 22. PMID 28012636
- [Background] Chu J, Duan W, Yu Z, Tao T, Xu J, Ma Q, Zhao L, Guo JJ. Intra-articular injections of platelet-rich plasma decrease pain and improve functional outcomes than sham saline in patients with knee osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2022 Dec;30(12):4063-4071. doi: 10.1007/s00167-022-06887-7. Epub 2022 Feb 6. PMID 35124707
- [Background] Nie LY, Zhao K, Ruan J, Xue J. Effectiveness of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Meta-analysis of Randomized Controlled Clinical Trials. Orthop J Sports Med. 2021 Mar 2;9(3):2325967120973284. doi: 10.1177/2325967120973284. eCollection 2021 Mar. PMID 33718505
- [Background] Singh H, Knapik DM, Polce EM, Eikani CK, Bjornstad AH, Gursoy S, Perry AK, Westrick JC, Yanke AB, Verma NN, Cole BJ, Chahla JA. Relative Efficacy of Intra-articular Injections in the Treatment of Knee Osteoarthritis: A Systematic Review and Network Meta-analysis. Am J Sports Med. 2022 Sep;50(11):3140-3148. doi: 10.1177/03635465211029659. Epub 2021 Aug 17. PMID 34403285
- [Background] Belk JW, Kraeutler MJ, Houck DA, Goodrich JA, Dragoo JL, McCarty EC. Platelet-Rich Plasma Versus Hyaluronic Acid for Knee Osteoarthritis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Am J Sports Med. 2021 Jan;49(1):249-260. doi: 10.1177/0363546520909397. Epub 2020 Apr 17. PMID 32302218
- [Background] Laudy AB, Bakker EW, Rekers M, Moen MH. Efficacy of platelet-rich plasma injections in osteoarthritis of the knee: a systematic review and meta-analysis. Br J Sports Med. 2015 May;49(10):657-72. doi: 10.1136/bjsports-2014-094036. Epub 2014 Nov 21. PMID 25416198
- [Background] O'Dowd A. Update on the Use of Platelet-Rich Plasma Injections in the Management of Musculoskeletal Injuries: A Systematic Review of Studies From 2014 to 2021. Orthop J Sports Med. 2022 Dec 9;10(12):23259671221140888. doi: 10.1177/23259671221140888. eCollection 2022 Dec. PMID 36532150
- [Background] Xiong Y, Gong C, Peng X, Liu X, Su X, Tao X, Li Y, Wen Y, Li W. Efficacy and safety of platelet-rich plasma injections for the treatment of osteoarthritis: a systematic review and meta-analysis of randomized controlled trials. Front Med (Lausanne). 2023 Jun 27;10:1204144. doi: 10.3389/fmed.2023.1204144. eCollection 2023. PMID 37441691